CLINICAL TRIAL: NCT05873010
Title: Effectiveness Of Manual Compression and Stretching for The Myofascial Trigger Points in Upper Trapezius and Levator Scapulae
Brief Title: Manual Compression and Stretching for The Myofascial Trigger Points in Upper Trapezius and Levator Scapulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/546
Record Dates: First submitted 2023-03-18; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual Compression and Stretching (Experimental)
  Interventions: Diagnostic Test: Manual Compression and Stretching

INTERVENTIONS:
Diagnostic Test: Manual Compression and Stretching — Manual Compression and Stretching for The Myofascial Trigger Points

SUMMARY:
To compare the effectiveness of manual compression and stretching for myofascial trigger points in upper trapezius and levator scapulae in male office workers

ELIGIBILITY:
Inclusion Criteria:

* male office workers with age of 25-45 working from Monday to Friday for 6-8 hours in a day.

Exclusion Criteria:

* male office workers having any past trauma, chronic illness, any recent surgery and systemic diseases.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
VAS (visual analogue scale) for pain | 6 Months
  Stretching for The Myofascial Trigger Points in Upper Trapezius and Levator Scapulae using VAS
mechanical algometer Scale for pain | 6 Months
  Stretching for The Myofascial Trigger Points in Upper Trapezius and Levator Scapulae using mechanical algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No